CLINICAL TRIAL: NCT05707598
Title: Multivisceral Radical Resection for Surgical T4b Colorectal Cancer: Propensity Score-matched Study Comparing the the Laparoscopic and Open Approaches
Acronym: C-PelvEx-01
Status: Completed | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jianqiang Tang, Associate professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC-2023
Record Dates: First submitted 2023-01-12; First posted 2023-02-01 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2023-02

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Multivisceral resection; Laparoscope
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Laparoscopic multivisceral resection group: Patients who underwent laparoscopic multivisceral resection for clinical T4b colorectal cancer
  Interventions: Procedure: Laparoscopic surgery
- Open multivisceral resection group: Patients who underwent open multivisceral resection for clinical T4b colorectal cancer

INTERVENTIONS:
Procedure: Laparoscopic surgery — The laparoscopic approach was used for the treatment of clinical T4b colorectal cancer
  Groups: Laparoscopic multivisceral resection group

SUMMARY:
This study attempts to compare safety and long-term oncological outcomes between laparoscopic surgery and open surgery in the treatment of clinical T4b Colorectal cancer.

DETAILED DESCRIPTION:
Laparoscopic surgery is controversial for patients with T4b colorectal cancer who require multivisceral resection. With the expansion of the indications for laparoscopic surgery in recent years, surgeons try to perform laparoscopic multivisceral resection for the treatment of clinical T4b colorectal cancer. In this study, investigators attempted to compare safety and long-term oncological outcomes between laparoscopic surgery and open surgery in the treatment of clinical T4b colorectal cancer.

This study was a multicenter retrospective cohort study based on a multicenter database which contained hospitalization. According to the operation method, the patients were divided into laparoscopic multivisceral resection group(patients who underwent laparoscopic surgery or conversion to open surgery) and open multivisceral resection group(patients who underwent open surgery directly). The short-term and long-term result was compared between groups.

ELIGIBILITY:
Inclusion Criteria:

1. The patient was pathologically diagnosed as colorectal adenocarcinoma by endoscopic biopsy before operation.
2. All patients were considered to have tumors invading adjacent organs after preoperative radiographic evaluation.
3. All patients were recommended to undergo radical surgery after preoperative multidisciplinary consultation.

Exclusion Criteria:

Patients with distant metastasis or recurrent colorectal cancer were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. The patients were diagnosed with colorectal cancer and the tumor was considered to have invaded the adjacent organs before surgery.
  2. The patient experienced multivisceral resection for surgical T4b colorectal cancer from January 2010 to December 2021.
  3. All of the operations were performed with either open or laparoscopic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 638 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
Blood loss | Until the end of the operation, an average of 8 hours.
  Blood loss is defined as intraoperative blood loss and measured in milliliters(ml).
Complications | Until the patient recovered and was discharged from the hospital, an average of 10 days.
  Complications are defined as all surgery-related adverse events postoperatively, such as anastomotic leak, infection, which are measured in frequency.
Hospital stay after surgery | Until the patient recovered and was discharged from the hospital, an average of 10 days.
  Hospital stay after surgery is defined as the length of time from the end of surgery to the discharge of patient, which is measured in days.

SECONDARY OUTCOMES:
Overall survival | The endpoint of the overall survival assessment is the last follow-up or patient death. Follow-up time is up to 72 months.
  Overall survival is defined as the time from the surgery to death or last follow-up, regardless of disease recurrence, which was measured in months.
Disease-free survival | The endpoint of the disease-free survival assessment is the last follow-up or disease recurrence. Follow-up time is up to 72 months.
  Disease-free survival is defined as the time from the surgery to disease recurrence or last follow-up, which was measured in months.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China